CLINICAL TRIAL: NCT04719793
Title: Umbilical Cord Derived Wharton's Jelly for Treatment of Knee Osteoarthritis
Brief Title: Umbilical Cord Derived Wharton's Jelly for Knee Osteoarthritis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: BioIntegrate (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIOINT - 2020UCWJ/knee OA
Record Dates: First submitted 2021-01-14; First posted 2021-01-22 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Osteoarthritis, Knee
Keywords: Knee Osteoarthritis; Umbilical Cord; Wharton's Jelly
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wharton's Jelly (Experimental): Intraarticular injection of Umbilical Cord-derived Wharton's Jelly
  Interventions: Biological: Umbilical Cord-derived Wharton's Jelly

INTERVENTIONS:
Biological: Umbilical Cord-derived Wharton's Jelly — Intraarticular injection

SUMMARY:
The purpose of this study is to determine the safety and efficacy of intraarticular injection of umbilical cord derived Wharton's Jelly for treatment of knee osteoarthritis symptoms.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common joint disorder in the United States (US), affecting approximately 12% (~30 million) of adults aged between 25 and 74 years. By 2030, the number of US adults with arthritis is expected to reach 67 million leading to continuous increase in number of total knee replacement surgeries. While total knee replacement surgeries have shown advantages, avoiding or delaying surgery appears desirable, both from medical and health care system perspective. Lowering the number of total knee replacement surgeries will also lead to a reduced number of costly revision surgeries. Published studies have also demonstrated that the outcomes after total knee replacement surgeries for patients with Grade II or III knee OA (on Kellgren-Lawrence scale) are worse compared to patients with Grade IV OA. Conventional treatment modalities including activity modification, physical therapy, pharmacological agents such as nonsteroidal anti-inflammatory drugs (NSAIDs), corticosteroids, viscosupplementation and narcotics have limitations and potential side effects. Thus, there is a need for alternative intervention for patients with Grade II or III knee OA.

Interest in the use of biologics for regenerative medicine applications has increased over the last decade. To be compliant in the United States (U.S.), biologics that adhere to the U.S. Food and Drug Administration (FDA) regulation of Human Cells, Tissues, and Cellular and Tissue-Based Products (HCT/P's) regulated under title 21, part 1271 of the Code of Federal Regulations (CFR) must meet all the conditions under section 361 of Public Health Safety (PHS) Act to be regulated solely under this section. According to this regulation, HCT/P's must meet the criteria of being minimally manipulated, for homologous use only, not to be combination products, to have no systemic effect, and to be non-dependent on the metabolic activity of the living cells. Despite increased use, there is insufficient literature assessing the amount of growth factors (GF), cytokines (CK), hyaluronic acid (HA) and extracellular vesicles (EV) including exosomes present in these products, and more specifically, umbilical cord derived Wharton's Jelly. In addition, there is limited or no literature assessing the safety and efficacy of umbilical cord derived Wharton's Jelly products via a clinical study.

To address the insufficient literature assessing the presence and quantity of GF, CK, HA and EV including exosomes, investigators formulated a novel umbilical cord derived Wharton's Jelly product and evaluated it for the presence of these factors. The results from this study demonstrated that the essential components of regenerative medicine, namely GF, CK, HA and EV, are all present in large quantities in the formulated Wharton's Jelly. This study was an essential preliminary step to better characterize this Wharton's Jelly formulation before performing clinical trials to determine safety and efficacy of this novel formulation for regenerative medicine applications.

The goal of the proposed study is to evaluate the safety and efficacy of intraarticular injection of umbilical cord derived Wharton's Jelly for treatment of knee osteoarthritis symptoms. Investigators also hypothesize that patients receiving intraarticular injection of Wharton's Jelly is safe and will show an improvement in their overall satisfaction, Numeric Pain rating Scale (NPRS), Knee Injury and Osteoarthritis Outcome Score (KOOS) and cartilage formation over a period of 1 year compared to the baseline visit.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 years or older.
2. Must have a body mass index (BMI) of < 40Kg/m2.
3. Must be able to comply with the requirements of study visits.
4. Diagnosed with mild to moderate knee osteoarthritis (OA) in one knee only - Grade 2 or 3 on the KL grading scale.
5. Pain score of 4 or more on the NPRS (on scale of 0 to 10).
6. Female patients were abstinent, surgically sterilized or postmenopausal.
7. Premenopausal females with negative pregnancy test, and who does not anticipate pregnancy and will actively practice an accepted contraceptive method for the duration of study.
8. Males with premenopausal female partners, will take contraceptive measures for the duration of study.
9. Be willing and capable of giving written informed consent to participate in this clinical study.
10. Be willing and capable of complying with study-related requirements, procedures and visits.

Exclusion Criteria:

1. Patients who have taken any pain medications including NSAIDs within 15 days (except Acetaminophen), prior to the study injection date, regularly use anticoagulants, substance abuse history, and/or failure to agree not to take any knee-symptom modifying drugs during the course of the study without discussing and reporting the use to site principal investigator and study team.
2. Patients who are positive on special tests and stability tests on the physical exam case report form.
3. Patients with intraarticular injection of any drug including corticosteroids, viscosupplementation in the index knee in last 3 months.
4. Patients with index knee surgery within last 6 months.
5. Patients with traumatic injury to index knee within last 3 months.
6. Patients with planned elective surgery during the course of the study.
7. Patients with organ or hematologic transplantation history, rheumatoid arthritis or other autoimmune disorders.
8. Patients on immunosuppressive medication/treatment, diagnosis of non-basal cell carcinoma within last 5 years.
9. Patients with knee infection or who used antibiotics for knee infection within last 3 months.
10. Patients who participated in another clinical trial or treatment with any investigational product within last 30 days prior to inclusion in the study.
11. Female patients who are breast feeding or are pregnant or desire to be pregnant during the course of the study.
12. Patients with contraindication to X-ray or MRI imaging.
13. Patients with serious neurological, psychological or psychiatric disorders.
14. Patients with other medical conditions determined by site principal investigator as interfering with the study.
15. Patients with an injury or disability claim under current litigation or pending or approved workers' compensation claim.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse effects as assessed by Comprehensive Metabolic Profile | 1week
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by Comprehensive metabolic profile
Treatment-emergent adverse effects as assessed by Comprehensive Metabolic Profile | 6weeks
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by Comprehensive metabolic profile
Treatment-emergent adverse effects as assessed by Comprehensive Metabolic Profile | 3months
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by Comprehensive metabolic profile
Treatment-emergent adverse effects as assessed by Comprehensive Metabolic Profile | 6months
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by Comprehensive metabolic profile
Treatment-emergent adverse effects as assessed by Comprehensive Metabolic Profile | 1year
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by Comprehensive metabolic profile
Treatment-emergent adverse effects as assessed by creatinine levels | 1week
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by creatinine levels
Treatment-emergent adverse effects as assessed by creatinine levels | 6weeks
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by creatinine levels
Treatment-emergent adverse effects as assessed by creatinine levels | 3months
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by creatinine levels
Treatment-emergent adverse effects as assessed by creatinine levels | 6months
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by creatinine levels
Treatment-emergent adverse effects as assessed by creatinine levels | 1year
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by creatinine levels
Treatment-emergent adverse effects as assessed by liver function tests | 1week
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by liver function tests
Treatment-emergent adverse effects as assessed by liver function tests | 6weeks
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by liver function tests
Treatment-emergent adverse effects as assessed by liver function tests | 3months
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by liver function tests
Treatment-emergent adverse effects as assessed by liver function tests | 6months
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by liver function tests
Treatment-emergent adverse effects as assessed by liver function tests | 1year
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by liver function tests
Treatment-emergent adverse effects as assessed by complete blood count | 1week
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by complete blood count
Treatment-emergent adverse effects as assessed by complete blood count | 6weeks
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by complete blood count
Treatment-emergent adverse effects as assessed by complete blood count | 3months
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by complete blood count
Treatment-emergent adverse effects as assessed by complete blood count | 6months
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by complete blood count
Treatment-emergent adverse effects as assessed by complete blood count | 1year
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by complete blood count
Treatment-emergent adverse effects as assessed by C-reactive protein | 1week
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by C-reactive protein
Treatment-emergent adverse effects as assessed by C-reactive protein | 6weeks
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by C-reactive protein
Treatment-emergent adverse effects as assessed by C-reactive protein | 3months
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by C-reactive protein
Treatment-emergent adverse effects as assessed by C-reactive protein | 6months
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by C-reactive protein
Treatment-emergent adverse effects as assessed by C-reactive protein | 1year
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by C-reactive protein
Treatment-emergent adverse effects as assessed by erythrocyte sedimentation rate | 1week
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by erythrocyte sedimentation rate
Treatment-emergent adverse effects as assessed by erythrocyte sedimentation rate | 6weeks
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by erythrocyte sedimentation rate
Treatment-emergent adverse effects as assessed by erythrocyte sedimentation rate | 3months
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by erythrocyte sedimentation rate
Treatment-emergent adverse effects as assessed by erythrocyte sedimentation rate | 6months
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by erythrocyte sedimentation rate
Treatment-emergent adverse effects as assessed by erythrocyte sedimentation rate | 1year
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by erythrocyte sedimentation rate
Treatment-emergent adverse effects as assessed by T, B and NK cell lymphocyte subsets | 1week
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by T, B and NK cell lymphocyte subsets
Treatment-emergent adverse effects as assessed by T, B and NK cell lymphocyte subsets | 6weeks
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by T, B and NK cell lymphocyte subsets
Treatment-emergent adverse effects as assessed by T, B and NK cell lymphocyte subsets | 3months
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by T, B and NK cell lymphocyte subsets
Treatment-emergent adverse effects as assessed by T, B and NK cell lymphocyte subsets | 6months
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by T, B and NK cell lymphocyte subsets
Treatment-emergent adverse effects as assessed by T, B and NK cell lymphocyte subsets | 1year
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by T, B and NK cell lymphocyte subsets
Treatment-emergent adverse effects as assessed by serum IgG, IgA, IgM and IgE levels | 1week
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by serum IgG, IgA, IgM and IgE levels
Treatment-emergent adverse effects as assessed by serum IgG, IgA, IgM and IgE levels | 6weeks
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by serum IgG, IgA, IgM and IgE levels
Treatment-emergent adverse effects as assessed by serum IgG, IgA, IgM and IgE levels | 3months
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by serum IgG, IgA, IgM and IgE levels
Treatment-emergent adverse effects as assessed by serum IgG, IgA, IgM and IgE levels | 6months
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by serum IgG, IgA, IgM and IgE levels
Treatment-emergent adverse effects as assessed by serum IgG, IgA, IgM and IgE levels | 1year
  To determine safety i.e. adverse events associated with intraarticular administration of Umbilical cord-derived Wharton's Jelly as assessed by serum IgG, IgA, IgM and IgE levels

SECONDARY OUTCOMES:
Change in patient reported outcome measures, Numeric Pain Rating Scale | Change from baseline to immediately after injection
  To determine change in patient reported outcome measure, Numeric Pain Rating Scale (NPRS). A decrease in score indicates improvement.
Change in patient reported outcome measures, Numeric Pain Rating Scale | Change from baseline to 24hours after injection
  To determine change in patient reported outcome measure, Numeric Pain Rating Scale (NPRS). A decrease in score indicates improvement.
Change in patient reported outcome measures, Numeric Pain Rating Scale | Change from baseline to 48hours after injection
  To determine change in patient reported outcome measure, Numeric Pain Rating Scale (NPRS). A decrease in score indicates improvement.
Change in patient reported outcome measures, Numeric Pain Rating Scale | Change from baseline to 1week after injection
  To determine change in patient reported outcome measure, Numeric Pain Rating Scale (NPRS). A decrease in score indicates improvement.
Change in patient reported outcome measures, Numeric Pain Rating Scale | Change from baseline to 6weeks after injection
  To determine change in patient reported outcome measure, Numeric Pain Rating Scale (NPRS). A decrease in score indicates improvement.
Change in patient reported outcome measures, Numeric Pain Rating Scale | Change from baseline to 3months after injection
  To determine change in patient reported outcome measure, Numeric Pain Rating Scale (NPRS). A decrease in score indicates improvement.
Change in patient reported outcome measures, Numeric Pain Rating Scale | Change from baseline to 6months after injection
  To determine change in patient reported outcome measure, Numeric Pain Rating Scale (NPRS). A decrease in score indicates improvement.
Change in patient reported outcome measures, Numeric Pain Rating Scale | Change from baseline to 1year after injection
  To determine change in patient reported outcome measure, Numeric Pain Rating Scale (NPRS). A decrease in score indicates improvement.
Change in patient reported outcome measures, Knee Injury and Osteoarthritis Outcome Score | Change from baseline to 1week after injection
  To determine change in patient reported outcome measure, Knee Injury and Osteoarthritis Outcome Score (KOOS). An increase in score indicates improvement.
Change in patient reported outcome measures, Knee Injury and Osteoarthritis Outcome Score | Change from baseline to 6weeks after injection
  To determine change in patient reported outcome measure, Knee Injury and Osteoarthritis Outcome Score (KOOS). An increase in score indicates improvement.
Change in patient reported outcome measures, Knee Injury and Osteoarthritis Outcome Score | Change from baseline to 3months after injection
  To determine change in patient reported outcome measure, Knee Injury and Osteoarthritis Outcome Score (KOOS). An increase in score indicates improvement.
Change in patient reported outcome measures, Knee Injury and Osteoarthritis Outcome Score | Change from baseline to 6months after injection
  To determine change in patient reported outcome measure, Knee Injury and Osteoarthritis Outcome Score (KOOS). An increase in score indicates improvement.
Change in patient reported outcome measures, Knee Injury and Osteoarthritis Outcome Score | Change from baseline to 1year after injection
  To determine change in patient reported outcome measure, Knee Injury and Osteoarthritis Outcome Score (KOOS). An increase in score indicates improvement.
Cartilage Formation | Change from baseline to 1year after injection
  To assess cartilage formation via MOCART (Magnetic Resonance Observation of Cartilage Repair Tissue). An increase in score indicates improvement.
Patient Satisfaction via 36-item short form survey (SF36) | Change from baseline to 3Months after injection
  To determine patient satisfaction via 36-item short form survey (SF36)
Patient Satisfaction via 36-item short form survey (SF36) | Change from baseline to 6Months after injection
  To determine patient satisfaction via 36-item short form survey (SF36)
Patient Satisfaction via 36-item short form survey (SF36) | Change from baseline to 1year after injection
  To determine patient satisfaction via 36-item short form survey (SF36)
Patient Satisfaction via 7-point Likert Scale | 1week after injection
  To determine patient satisfaction via 7-point Likert Scale. An increase in score indicates improvement.
Patient Satisfaction via 7-point Likert Scale | 6weeks after injection
  To determine patient satisfaction via 7-point Likert Scale. An increase in score indicates improvement.
Patient Satisfaction via 7-point Likert Scale | 3months after injection
  To determine patient satisfaction via 7-point Likert Scale. An increase in score indicates improvement.
Patient Satisfaction via 7-point Likert Scale | 6months after injection
  To determine patient satisfaction via 7-point Likert Scale. An increase in score indicates improvement.
Patient Satisfaction via 7-point Likert Scale | 1year after injection
  To determine patient satisfaction via 7-point Likert Scale. An increase in score indicates improvement.
Patient Satisfaction via Single Assessment Numeric Evaluation (SANE) | Change from baseline to 1week after injection
  To determine patient satisfaction via Single Assessment Numeric Evaluation (SANE). An increase in score indicates improvement.
Patient Satisfaction via Single Assessment Numeric Evaluation (SANE) | Change from baseline to 6weeks after injection
  To determine patient satisfaction via Single Assessment Numeric Evaluation (SANE). An increase in score indicates improvement.
Patient Satisfaction via Single Assessment Numeric Evaluation (SANE) | Change from baseline to 3months after injection
  To determine patient satisfaction via Single Assessment Numeric Evaluation (SANE). An increase in score indicates improvement.
Patient Satisfaction via Single Assessment Numeric Evaluation (SANE) | Change from baseline to 6months after injection
  To determine patient satisfaction via Single Assessment Numeric Evaluation (SANE). An increase in score indicates improvement.
Patient Satisfaction via Single Assessment Numeric Evaluation (SANE) | Change from baseline to 1year after injection
  To determine patient satisfaction via Single Assessment Numeric Evaluation (SANE). An increase in score indicates improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Saadiq F. El-Amin III, MD, PhD, Principal Investigator — El-Amin Orthopaedic & Sports Medicine Institute; Ashim Gupta, PhD, MBA, Study Director — BioIntegrate

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gupta A, Maffulli N, Rodriguez HC, Lee CE, Levy HJ, El-Amin SF 3rd. Umbilical cord-derived Wharton's jelly for treatment of knee osteoarthritis: study protocol for a non-randomized, open-label, multi-center trial. J Orthop Surg Res. 2021 Feb 18;16(1):143. doi: 10.1186/s13018-021-02300-0. PMID 33602286